CLINICAL TRIAL: NCT01556087
Title: Distress Tolerance and Reducing Early Relapse in Buprenorphine Patients
Brief Title: Distress Tolerance and Buprenorphine
Acronym: TRUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA032767
Record Dates: First submitted 2012-03-05; First posted 2012-03-16 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Opioid Dependence
Keywords: opioids; distress tolerance; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Distress Tolerance (Experimental): 7 sessions aimed at increasing distress tolerance skills
  Interventions: Behavioral: Distress Tolerance
- Health Education (Placebo Comparator): 7 didactic health education sessions
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Distress Tolerance — 7 individual sessions aimed at increasing distress tolerance skills
  Arms: Distress Tolerance
Behavioral: Health Education — 7 individual sessions with didactic health education information
  Arms: Health Education

SUMMARY:
The investigators propose that inability to tolerate the distress of opioid withdrawal and the negative affect associated with early abstinence are key factors in early illicit opioid lapse and subsequent buprenorphine treatment drop-out. Our intervention aimed at increasing distress tolerance is designed to increase treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* initiating buprenorphine treatment (which requires meeting current criteria for a DSM-IV diagnosis of opioid dependence)
* plan to remain on buprenorphine for at least three months
* age between 18 and 65 years
* if female of childbearing potential -- must be using adequate contraception (an intrauterine device, oral contraceptive, depot contraceptive, a barrier method "every time," or hysterectomy) as assessed by the study physician
* has at least two persons they regularly contact and can provide contact information for them
* speaks English sufficiently to understand instructions and assessments.

Exclusion Criteria:

* current methadone maintenance treatment program participation
* medically necessary prescription opioid treatment (e.g., for chronic pain)
* current criteria for a DSM-IV diagnosis of substance dependence for sedative/hypnotic drugs, alcohol, stimulants, cocaine, inhalants, hallucinogens
* a diagnosis of organic brain disorder, bipolar disorder, schizophrenia, schizo-affective, schizophreniform, or paranoid disorder, or major depression (subjects who meet criteria for "substance-induced mood disorder," or dysthymia only will not be excluded)
* current suicidality on the Modified Scale for Suicidal Ideation
* use of daily psychotropic, antidepressant, or anxiolytic medication
* evidence of neuropsychological dysfunction as assessed by the study physician with confirmation with the Folstein Mini-Mental Status Examination
* anticipated major painful event (significant surgical procedure) in the coming 6 months
* probation/parole requirements that might interfere with protocol participation
* history of allergic reaction to buprenorphine or naloxone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
the Client Satisfaction Questionnaire-8 | 4 months
  assess patient satisfaction with services
buprenorphine treatment adherence | 4 months
  adherence to buprenorphine treatment, which includes opioid use and risk behaviors, will be assessed

SECONDARY OUTCOMES:
distress tolerance persistence | 4 months
  mechanisms hypothesized to mediate the relationship between DT treatment and improved buprenorphine outcomes will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States